CLINICAL TRIAL: NCT04434872
Title: Fecal Microbiota Transplantation as a Treatment for Ulcerative Colitis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of budget
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0680-14-TLV
Record Dates: First submitted 2015-05-28; First posted 2020-06-17 (Actual); Last update posted 2020-06-17 (Actual); Status verified 2020-06

CONDITIONS: Ulcerative Colitis
Keywords: Microbiota; Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Colonoscopy; Gastroscopy; Fecal Microbiota Transplantation; Enema

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- FMT from a healthy donor (Active Comparator): Patients will undergo FMT 4 times during the study:
  first time, through a colonoscopy (sample volume: 250ml), and 3 more times (each sample volume: 100ml) during the following three days through:
  1. A Naso-jejunal feeding tube (that will be inserted through a gastroscopy) for patients suffering from colitis that involves more than 40 cm of the colon.
  2. Enemas, for patients suffering from colitis that involves the left colon up to 40 cm from the rectum.
  Interventions: Procedure: Colonoscopy; Procedure: Gastroscopy; Drug: Fecal Microbiota; Procedure: Enema
- FMT from a self donated stool sample (Placebo Comparator): Patients will undergo FMT 4 times during the study:
  first time, through a colonoscopy (sample volume: 250ml), and 3 more times (each sample volume: 100ml) during the following three days through:
  1. A Naso-jejunal feeding tube (that will be inserted through a gastroscopy) for patients suffering from colitis that involves more than 40 cm of the colon.
  2. Enemas, for patients suffering from colitis that involves the left colon up to 40 cm from the rectum.
  Interventions: Procedure: Colonoscopy; Procedure: Gastroscopy; Drug: Fecal Microbiota; Procedure: Enema

INTERVENTIONS:
Procedure: Colonoscopy — Fecal microbiota transplantation through colonoscopy
Procedure: Gastroscopy — Fecal microbiota transplantation through gastroscopy
Drug: Fecal Microbiota
Procedure: Enema — Fecal microbiota transplantation through enema

SUMMARY:
Ulcerative colitis (UC) is characterized by a disrupted homeostasis of the commensal bacterial population (dysbiosis). A promising therapy for restoration of the altered balance of the enteric microbiota is fecal microbial transplantation (FMT).

FMT will ameliorate colitis via alterations of patients' microbiota and their proteolytic-dependent effect on epithelial permeability.

Design: 80 patients will undergo 1:1 randomization for multiple FMT (Fecal Microbiota Transplantation) from a healthy donor or autologous (placebo) through colonoscopy and rectal enemas. The treating physicians and the patients will be blinded for the treatment arm.

At the FMT visit (first week), blood and stool samples will be taken and patients will be filling out questionnaires to assess disease activity level.

Every 2 weeks patients will come to a clinic for a follow up visit. 8 weeks after FMT, patients will undergo sigmoidoscopy to assess disease severity, biopsies will be taken as well.

ELIGIBILITY:
Inclusion Criteria:

* Over 3 month diagnosis of ulcerative colitis
* Active Colitis disease with endoscopic score >0
* Ability to sign an informed consent

Exclusion Criteria:

* Acute neutrophilia (under 500 neutrophils)
* Clostridium difficile infection
* Exposure to antibiotics 2 weeks prior to enrollment.
* Severe immune deficiency
* Hospitalization
* Proctitis involving less than 10cm of the rectum
* Malignancy with the past 5 years (excluding BCC)
* An unstable dose of steroids or 5ASA (5- aminosalicylic acid) with the past 2 weeks or of immunomodulators or biologic therapy within the past 12 weeks

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2015-07; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Clinical improvement | 8 weeks after FMT
  A composite measure- Will be measured by SCCAI (Simple Clinical Colitis Activity Index) and by MAYO SCORE

SECONDARY OUTCOMES:
Histological remission assessed by sigmoidoscopy | 8 weeks after FMT
  Will be assessed by sigmoidoscopy
Long term remission assessed through questionnaires | one year after FMT
  Will be assessed through questionnaires

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Gastroentherology, Tel Aviv, Israel